CLINICAL TRIAL: NCT01993732
Title: Ovarian Tissue Cryopreservation As A Means Of Preserving Ovarian Function in Females Undergoing Therapeutic Procedures That Will Potentially Lead To The Irreversible Loss of Ovarian Function
Brief Title: Ovarian Tissue Cryopreservation in Females Undergoing Procedures That Will Potentially Lead To Loss of Ovarian Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Estil Strawn, Professor, Director of Division of Reproductive Endocrinology and Infertility, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 126204
Record Dates: First submitted 2013-09-18; First posted 2013-11-25 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Cancer; Effects of Chemotherapy; Unspecified Complication of Bone Marrow Transplant; Auto Immune Disease
Keywords: Cancer; Cryopreservation; Ovarian Function; In Vitro
MeSH Terms: conditions — Neoplasms | interventions — Cryopreservation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Retrieval and Cryopreservation (Experimental): Females undergoing therapeutic procedures that will potentially lead to the irreversible loss of ovarian function will have their ovarian tissue retrieved and cryopreserved. Ideally, after treatment, the cryopreserved ovarian tissue can be thawed and auto-transplanted and ovarian function resumed.
  Interventions: Procedure: Retrieval and Cryopreservation

INTERVENTIONS:
Procedure: Retrieval and Cryopreservation — Females undergoing therapeutic procedures that will potentially lead to the irreversible loss of ovarian function will have their ovarian tissue retrieved and cryopreserved. Ideally, after treatment, the cryopreserved ovarian tissue can be thawed and auto-transplanted and ovarian function resumed.

SUMMARY:
The purpose of this study is to retrieve and cryopreserve ovarian tissue from females undergoing a treatment that may lead to irreversible loss of ovarian function.

DETAILED DESCRIPTION:
The aim of this preliminary study is to retrieve and properly cryopreserve ovarian tissue for autotransplantation in any premenopausal female whose ovarian function is threatened in a physiological, pathological or iatrogenic manner in an effort to observe the return of ovarian endocrine function and development of egg(s) appropriate for use in in vitro fertilization.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be female.
* Patient must have a disease process where the disease or its treatment adversely affects ovarian function.
* Patient must be recommended for this study by their oncologist or specialist.
* Patient (or legally authorized representative) must sign an informed consent.

Exclusion Criteria:

* Patients cannot be male.
* Patients must not be HIV positive.
* Patient cannot have a poor diagnosis such that she is not expected to survive to adulthood.
* Patient cannot have any medical condition that would contraindicate surgery.
* Patient cannot have any medical condition that would contraindicate general anesthesia.
* Patient cannot have any medical condition that would contraindicate pregnancy.

Min Age: 3 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-08-06 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Return of hormones produced by the ovarian tissue | 3 months after re-implantation

SECONDARY OUTCOMES:
Development of egg(s) appropriate for use in in vitro fertilization | Participants will be followed through their reproductive years (until the patient reaches 45 years of age)

CONTACTS AND LOCATIONS:
Overall Officials: Estil Strawn, MD, Principal Investigator — Medical College of Wisconsin
Locations (2):
- United States (2):
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
  - Froedtert and The Medical College of Wisconsin, Milwaukee, Wisconsin